CLINICAL TRIAL: NCT07395544
Title: Gait Training for Hemiplegic Stroke Patients: Employing a Stationary Neuro-developmental Trainer With Auditory Cues
Brief Title: Gait Training for Hemiplegic Stroke Patients With Stationary Trainer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHGH-(1069)112A-60
Record Dates: First submitted 2025-07-17; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: In this study, inertial measurement units are used for gait phase detection and as feedback parameters for the system. Previous studies have validated the reliability and accuracy of IMU data compared to those collected in motion analysis laboratories.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NDT gait training group (Experimental): NDT gait trainer which can automatically repeat NDT intervention, thereby alleviating therapists' workload and extending patients' training time. They analyzed therapists' intervention in manual NDT training and concluded that therapists cued subjects' anterior superior iliac spines (ASISs) when perceiving opposite heel strikes (HSs).
  Interventions: Device: NDT Gait Training System

INTERVENTIONS:
Device: NDT Gait Training System — The intervention includes a NDT gait training device that mimics therapist techniques through mechanical assistance, synchronized with auditory feedback and real-time gait analysis using IMU sensors.

SUMMARY:
This study aims to evaluate the effectiveness of a novel mobile neurodevelopmental treatment (NDT) gait training device for patients recovering from stroke. Stroke is a major cause of disability worldwide, and many survivors experience difficulty with walking and require long-term rehabilitation. NDT is a widely used rehabilitation approach that focuses on improving motor control through techniques such as facilitation, inhibition, and key point control. However, traditional NDT gait training can be physically demanding for therapists and often limits the training intensity and duration for patients.

To address these challenges, this study introduces an automated NDT gait training device that replicates therapist techniques using mechanical support and sensory feedback. The system uses bilateral dynamic assistance at the waist, auditory cues, and wearable inertial measurement units (IMUs) to help patients practice natural and symmetric walking patterns on the ground, instead of being restricted to treadmill training. The IMUs also provide objective gait data to assess improvement in gait symmetry, pelvic rotation, walking speed, and cadence.

The primary goal is to assess changes in these gait parameters before and after NDT-based intervention. The study plans to enroll 40 adult stroke survivors (aged 20 and older) over a 3-year period starting from May 1, 2024.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years, first-ever stroke, with Brunnstrom stage III to IV of the affected lower limb motor recovery.
* Functional Ambulation Category (FAC) level IV.
* Ability to ambulate on level ground without assistive devices.
* Ability to understand instructions and cooperate with assessments.

Exclusion Criteria:

* Presence of severe spinal cord injury or peripheral neuropathy.
* Unstable gait requiring assistive devices, or participants at high risk of falling.
* Severe impairment in vision, hearing, or cognition, making them unable to comply with assessments.
* Lower limb fracture within the past 6 months.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pelvic rotation | Baseline (pre-intervention) and post-intervention (immediately after completion of the NDT gait training program).
  The gait parameter will be collected using wearable inertial measurement units (IMUs) before and after the NDT gait training intervention and pelvic rotation will be measured through axial angular velocity
Walking speed | Baseline (pre-intervention) and post-intervention (immediately after completion of the NDT gait training program).
  Walking speed will be estimated from IMU during walking and reported in meters per second (m/s).
Step length | Baseline (pre-intervention) and post-intervention (immediately after completion of the NDT gait training intervention).
  Step length will be derived from IMU-based spatiotemporal gait data collected during overground walking and reported in meters (m).

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Fu Chen, MD, PhD, Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Beitou Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No